CLINICAL TRIAL: NCT03041857
Title: Understanding GMK Sphere Implant Tibiofemoral Kinematics by Means of Dynamic Videofluoroscopy
Status: Completed | Type: Observational
Sponsor: Dr. Renate List (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); Balgrist University Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Renate List, Doctor of Sciences (Dr. sc. ETH), Institute for Biomechanics, ETH Zürich
Organization: Institute for Biomechanics, ETH Zürich (Other)
Other Study IDs: MedactaGMKSphere
Record Dates: First submitted 2016-03-04; First posted 2017-02-03 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Total Knee Arthroplasty; Tibiofemoral Kinematics
Keywords: Videofluoroscopy; GMK Sphere; GMK PS Fixed Bearing; GMK UC Mobile Bearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GMK Sphere: Subjects with a unilateral Medacta GMK Sphere TKA
  Interventions: Radiation: Observational use of fluoroscopy
- GMK PS: Subjects with a unilateral Medacta GMK Primary PS Fixed Bearing TKA
  Interventions: Radiation: Observational use of fluoroscopy
- GMK UC: Subjects with a unilateral Medacta GMK Primary UC Fixed Bearing TKA
  Interventions: Radiation: Observational use of fluoroscopy

INTERVENTIONS:
Radiation: Observational use of fluoroscopy

SUMMARY:
The objective of this research project is to perform a comparative study on the in vivo kinematics of the GMK Sphere prosthesis in comparison to the conventional GMK PS Fixed Bearing TKA as well as to the GMK UC Mobile Bearing during level walking, stair descent and downhill walking by means of videofluoroscopy.

DETAILED DESCRIPTION:
Total arthroplasty of the knee (TKA) aims to relieve patient pain and improve functionality of the joint. To maintain sufficient range of motion, but also not overload the surrounding soft tissue structures, reproduction of tibio-femoral kinematics of the healthy knee is thought to be beneficial. In previous studies, it has been shown that the medial condyle, described by the centre of the medial condylar sphere, does not move anterioposteriorly during progressing joint flexion, whereas the lateral condyle has been observed to translate in a posterior direction producing tibial internal rotation with flexion (Freeman and Pinskerova 2003, Pinskerova, Johal et al. 2004, Freeman and Pinskerova 2005). The GMK Sphere prosthesis is specifically designed to mimic the healthy kinematics with providing a medial pivot.

The objective of this research project is to perform a comparative study on the in vivo kinematics of the GMK Sphere prosthesis in comparison to the conventional GMK PS Fixed Bearing TKA as well as to the GMK UC Fixed Bearing. The study includes the simultaneous assessment of the 3D kinematics of the TKA by means of an automated moving fluoroscope and subsequent 2D/3D registration based on CAD models of the TKA, whole leg kinematics by means of skin markers and ground reaction forces during level walking, stair descent and downhill walking a 10° inclined slope. Precisely, the aim is to assess tibio-femoral kinematics in 8-10 TKA subjects implanted one or more years previously with the GMK Sphere prosthesis. In addition, 8-10 conventional GMK PS Fixed Bearing TKA subjects, as well as 8-10 GMK UC Mobile Bearing TKA subjects will be measured to provide a comparison against the GMK Sphere prosthesis kinematics.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age: 40 to 100 years
* Unilateral TKA
* ≥ 1 years postoperatively
* BMI ≤ 33
* Good outcome, WOMAC between 0 to 28 (0-14 (Excellent), 15-28 (Good)) No pain subjects, VAS ≤ 2
* Good health condition, adequate for test procedure

Exclusion Criteria:

* Other actual significant problem on lower extremities
* Any other arthroplasty at the lower extremities
* Subject incapable to understand and sign informed consent
* Pregnancy at time of testing
* Incapable of performing the motion tasks
* Misaligned TKA (≥ ± 3° from mechanical axis)

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants fulfilling all of the following inclusion criteria are eligible for the study. The presence of any one of the following exclusion criteria will lead to the exclusion of the participant.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the three-dimensional kinematics of the GMK Sphere Fixed Bearing TKA to the kinematics of the GMK Primary PS fixed bearing and GMK Primary UC Mobile Bearing TKA. | 3 hours
  With video-fluoroscopic assessment it is possible to directly measure the kinematics of the tibial and the femoral components in vivo during daily activities, such as level walking, downhill walking and stair descent. Thus, for the first time the present study provides in vivo assessed data of the 3D motion of the GMK Sphere System during daily activities. The knowledge of the in vivo kinematic behaviour of the GMK Sphere System compared to conventional GMK PS Fixed Bearing and GMK UC Mobile Bearing TKA leads to an improved understanding of the design principle. Observation of the kinematics in terms of range of motion, patterns of anterior-posterior motion of medial and lateral condyle points ("posterior femoral rollback") and tibio-femoral internal/external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Renate List, Dr., Principal Investigator — Institute for Biomechanics, ETH Zurich
Locations (1):
- Institute for Biomechanics, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No